CLINICAL TRIAL: NCT02180425
Title: The Lipid Profile of the Skin Surface in Acne
Acronym: Acne
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 531506
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Acne
Keywords: acne; lipid; tretinoin; isotretinoin
MeSH Terms: conditions — Acne Vulgaris | interventions — Tretinoin; Adapalene; Isotretinoin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sebum collections from sebutapes
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Healthy Group: The subjects in this group do not have a history of acne.
- Acne Group, Topical Retinoid: These subjects have been prescribed a topical retinoid for their acne. They will participate in the study for a period of 1 month.
  Interventions: Drug: Tretinoin or Adapalene
- Acne Group, Isotretinoin: These subjects have been prescribed isotretinoin for their acne. They will participate in the study for a period of 5-6 months.
  Interventions: Drug: Isotretinoin

INTERVENTIONS:
Drug: Tretinoin or Adapalene — Subjects will apply a pea sized amount of topical retinoid cream once daily at night for 30 days. Subjects will return for a follow-up visit.
  Other Names: Retin A
  Groups: Acne Group, Topical Retinoid
Drug: Isotretinoin — Subjects will take one pill once daily for 5 months. Subjects will return after 1 month and after 4-5 months of treatment for skin lipid profiling.
  Other Names: Accutane
  Groups: Acne Group, Isotretinoin

SUMMARY:
The purpose of this study is to evaluate the differences in the skin lipid profile of patients with and without acne. Secondly, the goal is to learn more about what the effects of retinoinds (topical and systemic) are on the the skin lipid profile. We hypothesize that the skin lipid profile of subjects with acne will be lower in inflammatory lipids in comparison to subjects without acne.

DETAILED DESCRIPTION:
Skin lipid profile will be conducted via sebutapes- adhesive tapes that painlessly absorbs sebum from the face. These tapes will be placed on the face for 1 hour. A photograph of the face will be taken during each study visit. A sebumeter will also be used to measure skin sebum secretion rate.

ELIGIBILITY:
Inclusion Criteria:

* age 12 to 30 years
* have been prescribed tretinoin OR isotretinoin

Exclusion Criteria:

* those who have taken isotretinoin (systemic)
* those who used tretinoin or other topical retinoid within two weeks of starting the study
* those with seborrheic dermatitis, rosacea, or polycystic ovary syndrome
* those who are pregnant, prisoners, or cognitively impaired
* those who do not fit the inclusion criteria

Ages: 12 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Subjects will be from the UC Davis Dermatology Clinic, surrounding dermatology clinics, from the UC Davis undergraduate campus, and from the California State University Sacramento campus.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Skin lipid profile of acne and healthy patients | baseline visit
  Compare the skin lipid profile of acne and healthy patients at baseline

SECONDARY OUTCOMES:
Skin lipid profile of acne patients after treatment | at 1 month and 4-5 months of treatment
  Patients in the topical retinoid group will have their lipids evaluated after 1 month of treatment. Patients in the systemic retinoid (isotretinoin) group will have their lipids evaluated after 1 and 4-5 months of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Raja K Sivamani, MD, Principal Investigator — UC Davis
Locations (2):
- United States (2):
  - Dermatology Research Area, Davis, California
  - UC Davis Department of Dermatology, Sacramento, California

REFERENCES:
- [Background] Thody AJ, Shuster S. Control and function of sebaceous glands. Physiol Rev. 1989 Apr;69(2):383-416. doi: 10.1152/physrev.1989.69.2.383. PMID 2648418
- [Background] Blume U, Verschoore M, Poncet M, Czernielewski J, Orfanos CE, Schaefer H. The vellus hair follicle in acne: hair growth and sebum excretion. Br J Dermatol. 1993 Jul;129(1):23-7. doi: 10.1111/j.1365-2133.1993.tb03306.x. PMID 8369207
- [Background] Zouboulis CC, Baron JM, Bohm M, Kippenberger S, Kurzen H, Reichrath J, Thielitz A. Frontiers in sebaceous gland biology and pathology. Exp Dermatol. 2008 Jun;17(6):542-51. doi: 10.1111/j.1600-0625.2008.00725.x. PMID 18474083
- [Background] Doshi A, Zaheer A, Stiller MJ. A comparison of current acne grading systems and proposal of a novel system. Int J Dermatol. 1997 Jun;36(6):416-8. doi: 10.1046/j.1365-4362.1997.00099.x. No abstract available. PMID 9248884
- [Background] Morello AM, Downing DT, Strauss JS. Octadecadienoic acids in the skin surface lipids of acne patients and normal subjects. J Invest Dermatol. 1976 May;66(5):319-23. doi: 10.1111/1523-1747.ep12482300. PMID 131844
- See also: University of California-Davis Department of Dermatology Clinical Research — http://www.ucdmc.ucdavis.edu/dermatology/research/clinical